CLINICAL TRIAL: NCT02799732
Title: A Feasibility Study for the Clinical Trial: "A Scientific Evaluation of One and Two Doses of the Bivalent and Nonavalent Prophylactic HPV Vaccines" (1DT)
Brief Title: A Feasibility Study for the One-dose Clinical Trial (1DT)
Acronym: FS-ESCUDDO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundación Inciensa (Other)
Responsible Party: Principal Investigator, Paula Gonzalez Maya, Director and Investigator, Fundación Inciensa
Other Study IDs: CEC-ICIC-E085-2016
Record Dates: First submitted 2016-05-30; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Compliance
Keywords: Feasibility Study; HPV vaccine; 1Dose Trial
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — De-identified samples will be retained to be used as controls in the main trial.
Oversight: Data Monitoring Committee: No

SUMMARY:
This feasibility study was developed to evaluate the proposed approaches for enrollment, sample collection, interview and retention over a six-month vaccination period for the clinical trial: "A scientific evaluation of one and two doses of the bivalent and nonavalent prophylactic HPV vaccines" (1DT) currently under development . These aspects will be assessed quantitatively and qualitatively by measuring the efforts needed to identify and recruit each study participant, the participation rate for the study, and the retention rate at six months, as well as collecting information on the acceptability of study procedures. To supplement the assessment of the acceptability of the self-collected swab among older girls, a parallel effort will be done at the end of this feasibility study. Combined, this feasibility work will allow for modifications to the design, approaches and methods of the new trial.

DETAILED DESCRIPTION:
Selection of study population and recruitment. Costa Rica is divided in provinces that are further divided in cantons, which are subdivided into districts. Districts are conceptually divided into minimal geo-statistical units (MGUs), territorial units roughly equivalent to a block. These MGUs were defined by the National Institute of Statistics and Census (INEC) for the national census conducted in 2011; digital maps and census data by age and gender for MGUs are available.

The study area being proposed for the 1DT was defined to reach an adequate catchment area in order to fulfill 1DT enrollment goals of 20,000 girls. This defined area includes ~125,000 girls in regions where previous NCI/PEG studies were conducted as well as new provinces.

For the feasibility study, three urban and three rural districts from three different provinces were selected: San Ignacio de Acosta and Tibas in San José; Desamparados and Cirri Sur in Alajuela and, Liberia and San Antonio de Nicoya in Guanacaste. MGUs in these districts will be ordered randomly and the first MGU within the selection will visited. An experienced study outreach worker (OW) will visit all houses within the selected MGU and will enumerate and collect information on all girls ages 12 to 16 residing in the MGU. At that time, if a potentially-eligible girl is present, the OW will invite her to participate in the feasibility study by informing her and her parent/legal guardian of the feasibility study, and if interested, will assign a participant study ID (PID). The informed consent/assent process for the feasibility study will be conducted at that time. Once consented/assented, the girl will be appointed to a medical office close to her house, where she will be expected to attend the feasibility study visit. If a potential participant or her parent/legal guardian is not present, the OW will leave study materials with the household and arrange to return at another time to discuss the study. The brochure will include a phone number in case the girl/parents want to get additional information by phone. Within an MGU, five contact attempts will be made per house. Once all houses in the selected MGU have been visited, if fewer than 15 households of participants have been enrolled, the next random selected MGUs will be visited (note, this is defined as girls in a household instead of individuals girls since girls within a household will likely be correlated in their response rate). If 15 or more households of participants have been enrolled after visiting the originally-selected MGU, then the team will move to the next district. This procedure will be repeated until approximately 15 girls have been enrolled in the district, but once an MGU is selected and visited, all houses in that MGU should be visited before moving to another district, even if more than 15 girls are enrolled, to allow for valid computation of the participation rate.

Data on the number of houses approached, average number of visits necessary to collect information in each house (maximum of five visits), percentage of houses contacted during first visit, subsequent visits, number of houses where it was not possible to obtain information, number with girls in the age range, number of girls potentially eligible as determined during home visit, number which consent and agree to attend a study visit, and the true number of girls who attend the study visit, will be collected.

Feasibility Study Clinic Visits. The guiding principle for the feasibility clinic visit is that it should parallel the clinic visits planned for the 1DT up to the point of randomization (which cannot be mocked in the feasibility study).

Consent/assent/enrolment medical history. The first feasibility study clinic visit will start with an explanation of the proposed informed consent and assent of the 1DT (in other words, a mock consent procedure). Girls will be asked if they would be willing to participate in such study. A clinician will then obtain a medical history from the girl and her parent/legal guardians and, if the medical doctor considers necessary based on the medical history, she will perform a physical examination to confirm good general health. Reproductive history and hormonal contraceptive use will also be obtained by the doctor.

Questionnaire. A self-administered questionnaire will then be administered. It will query information on years of education, socio-economic status, menstrual history, sexual history, and smoking. The questionnaire will be used to evaluate acceptance of self-administered questionnaire, perception of the sense of confidentiality of the answers provided, ability to understand the questions, percentage of girls needing help and completeness of the responses. Girls will be also presented with a picture of the female genital anatomy in order to evaluate their capacity to identify where a self-collected swab should be inserted.

Urine. In the 1DT, all participants will be asked to collect 15mL urine specimens for a urine pregnancy test and to store residual volume for HPV testing. While we are not conducting the pregnancy test or the HPV testing during this feasibility study, we aim to evaluate the acceptability of collecting urine following the specific procedure needed to obtain urine samples suitable for HPV testing.

Spit. In the 1DT, the immunogenicity subcohort will be asked to provide a saliva sample by spitting into a cryovial using a straw for the evaluation of mucosal immune response. Thus, we plan to investigate the acceptability of this sample.

Blood. In the 1DT, blood specimens will be collected from all participants at the two vaccination visits, the twelve-month visit and yearly after that. The purpose of these blood collections will be to monitor immune response to vaccination. We will ask participants in the feasibility study to provide a total of 10 mL of blood. To assure that participation and retention rates in our trial are not negatively affected by the blood draws, refusal to have blood collected will be allowed, and will be documented.

Self-collected Cervicovaginal Sample. In the 1DT, self-collected cervicovaginal samples will be used for HPV testing. Participants 15 and older who report having had sexual intercourse will be asked to self-collect a cervicovaginal sample.

In order to protect participant confidentiality, study staff will administer detailed instructions and materials for sample collection to all participants 15 and older irrespective of sexual experience. All these participants will be instructed to collect the sample only if appropriate (defined as being sexually active). Refusal to collect this specimen among sexually-active girls will be documented. The self-collected cervicovaginal samples collected as part of the feasibility study will be used to assess the adequacy of the sample.

Participants will be asked about their impressions of the study procedures and time expended. At the conclusion of the visit, they will receive a voucher for HPV vaccination at a local pharmacy, while in the 1DT, vaccination would be offered during the study visit.

Six-month feasibility study visit. The second visit will occur six months following the baseline study visit. Qualified staff will conduct the second feasibility study visit, which will include a self-administered questionnaire addressing behaviors during the time between the enrollment and six-month study visit, blood specimen collection, and among participants age 15 and older who report having had sexual intercourse, a self-collected cervicovaginal sample. After answering questions about their impressions on the second visit procedures, they will receive a voucher for the second dose of the vaccine.

Biological specimens obtained from participants in this study will be processed and stored to evaluate quality of the sample and to generate de-identified pools of specimens to be used as quality control specimens for various assays planned as part of the overall planning for the One-dose trial. This could allow for the formal evaluation of assay performance and testing batch effects in our future testing and maximize the quality of the research we conduct.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent must be able to communicate with study staff
* Must live in the study area
* Must sign Informed Assent
* Parent must sign Informed Consent
* Adolescent must be in good general health

Exclusion Criteria:

-Planning to move out of study area in the following 6 months

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescent girls aged 12 to 16 living in rural and urban areas of three Costa Rican provinces, included in the geographical areas considered for inclusion in the IDT.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled per total inhabitants in same age range in study area | 11 months
  Estimated response rate among girls aged 12 to 16 residing in rural and urban areas of three Costa Rican provinces considered for inclusion in the 1DT, which will be computed as the number of girls who come to a study clinic and complete the mock consent of the IDT divided by the number of estimated girls in the age range on the 2011 Costa Rican national census.

SECONDARY OUTCOMES:
Number of houses canvassed per registered adolescents | 11 months
  Quantify the field effort (amount of houses canvassed in census) required to identify and contact each potentially eligible participant
Number of participants completing second study visit per total of study participants | 11 months
  Determine retention rates of participation at 6 months

IPD SHARING:
Plan to Share IPD: No